CLINICAL TRIAL: NCT05260008
Title: A Phase 2B, Randomized, Double Blind, Active Comparator, Multicenter, Safety, and Efficacy Trial of ATX-101 in Subjects Undergoing Total Knee Arthroplasty
Brief Title: Study Assessing Pain Relief After Replacement of the Knee
Acronym: SPARK
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Based on positive data from the dose-ranging portion of the study, Sponsor decided as of May 28, 2024 not to move forward with the previously designed global ATX101-TKA-003 study.
Sponsor: Allay Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ATX-101-TKA-003
Record Dates: First submitted 2022-02-18; First posted 2022-03-02 (Actual); Results first posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-07

CONDITIONS: Acute Postoperative Pain
Keywords: postoperative pain; post-surgical pain total knee arthroplasty; total knee replacement ATX-101; bupivacaine; bupivacaine implant
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine; Epinephrine

STUDY DESIGN:
Intervention Model Description: This is a Phase 2B, randomized, double blind, active comparator multicenter trial in participants undergoing total knee arthroplasty.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- ATX-101 Dose A (Experimental): ATX-101 Dose A
  Interventions: Drug: ATX-101
- ATX-101 Dose B (Experimental): ATX-101 Dose B
  Interventions: Drug: ATX-101
- bupivacaine hydrochloride (Active Comparator): bupivacaine hydrochloride without epinephrine via local infiltration and/or nerve block
  Interventions: Drug: bupivacaine hydrochloride without epinephrine

INTERVENTIONS:
Drug: ATX-101 — ATX-101 (bupivacaine) implant, one-time administration into the surgical site
  Arms: ATX-101 Dose A
Drug: ATX-101 — ATX-101 (bupivacaine) implant, one-time administration into the surgical site
  Arms: ATX-101 Dose B
Drug: bupivacaine hydrochloride without epinephrine — bupivacaine hydrochloride (125 mg) without epinephrine via local infiltration and/or nerve block
  Arms: bupivacaine hydrochloride

SUMMARY:
This is a Phase 2B randomized, double blind, active controlled, multi-center clinical trial to evaluate the safety and efficacy of ATX-101 in participants following total knee arthroplasty. The following is short title and acronym for the study: Study Assessing Pain Relief after Replacement of the Knee (SPARK)

ELIGIBILITY:
Inclusion Criteria:

* Primary indication of total knee arthroplasty is knee pain due to osteoarthritis or post-traumatic arthritis.
* Scheduled to undergo primary unilateral total knee arthroplasty with a cemented prosthesis, without use of a surgical drain, and under bupivacaine spinal anesthesia (dextrose is permitted).
* American Society of Anesthesiology (ASA) Physical Classification System of class 1, 2 or 3.

Exclusion Criteria:

* Has a planned concurrent surgical procedure.
* Has had any previous arthroplasty, unicompartmental knee arthroplasty or total knee arthroplasty in the study knee or previous arthroplasty, unicompartmental knee arthroplasty, or total knee arthroplasty in the contralateral knee within 6 months prior to screening.
* Has been administered any type of intra-articular injection within 3 months of surgery in the trial knee.
* Immunocompromised or has a known history of Hepatitis B, human immunodeficiency virus (HIV), or Hepatitis C.
* Routinely take opioid analgesics and are expected to require opioid analgesics in the postsurgical period that is not strictly related to the trial.
* Unable to abstain from opioid use for knee pain within 14 days of surgery.
* Has been administered systemic steroids within 14 days prior to surgery.
* Has been administered any local anesthetic within 5 days prior to the scheduled surgery.
* Screening electrocardiogram (ECG) with significant abnormalities associated with significant heart disease.
* Has a contraindication or a known suspected history of allergy, hypersensitivity or idiosyncratic reaction to trial medications.
* Has uncontrolled depression, anxiety, psychiatric, or neurological disorder that might interfere with trial study assessments.
* Has a medical condition or receiving medication such that, in the opinion of the investigator, participating in the trial would pose a health risk to the subject or might interfere with the study outcome.
* Has a known or suspected history of drug or alcohol abuse. A subject with a history of alcohol use disorder that has ≥10 years sobriety will be permitted.
* Has received/used an investigational drug, product, or device for a clinical trial within 30 days of screening. COVID-19 vaccines are permitted if the subject is not in a clinical trial for the vaccine.
* Has a Body Mass Index (BMI) ≥45 kg/m2

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2022-06-07 (Actual); Primary Completion 2024-01-15 (Actual); Study Completion 2024-01-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (13):
- Australia (5):
  - Prince of Wales Private Hospital, Sydney, New South Wales
  - John Flynn Private Hospital, Tugun, Queensland
  - Royal Adelaide Hospital / PARC Clinical Research, Adelaide, South Australia
  - St Andrew's Private Hospital, Adelaide, South Australia
  - The Avenue Private Hospital, Windsor, Victoria
- Canada (2):
  - Durham Bone and Joint Specialists, Ajax, Ontario
  - London Health Sciences Centre - University Hospital, London, Ontario
- United Kingdom (6):
  - Department of Trauma and Orthopaedic Surgery, Addenbrooke's Hospital, Cambridge, Cambridgeshire
  - Southampton General Hospital, Southampton, Hampshire
  - Royal National Orthopaedic Hospital, Stanmore, Middlesex
  - Nottingham Elective Orthopaedic Service, Nottingham University Hospitals, Nottingham, Nottinghamshire
  - Robert Jones & Agnes Hunt Orthopaedic Hospital, Oswestry, Shropshire
  - Chapel Allerton Hospital C/O The Leeds Teaching Hospitals NHS Trust, Leeds, West Yorkshire

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- ATX-101 1000 mg: ATX-101 1000 mg
  ATX-101: ATX-101 (bupivacaine) implant, one-time administration into the surgical site
- ATX-101 1500 mg: ATX-101 1500 mg
  ATX-101: ATX-101 (bupivacaine) implant, one-time administration into the surgical site
- Bupivacaine Hydrochloride: bupivacaine hydrochloride
  bupivacaine hydrochloride without epinephrine via local infiltration and/or nerve block
- Saline Placebo: Saline Placebo
  saline placebo (0.9%) sodium chloride via local infiltration
Period: Overall Study
Arm/Group | ATX-101 1000 mg | ATX-101 1500 mg | Bupivacaine Hydrochloride | Saline Placebo
Started | 37 | 37 | 34 | 4
Completed | 37 | 36 | 34 | 4
Not Completed | 0 | 1 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ATX-101 1000 mg | ATX-101 1500 mg | Bupivacaine Hydrochloride | Saline Placebo | Total
Number analyzed (Participants) | 37 | 37 | 34 | 4 | 112
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 15 | 15 | 14 | 2 | 46
  >=65 years | 22 | 22 | 20 | 2 | 66
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.2 (8.12) | 68.3 (6.89) | 67.5 (7.62) | 63.0 (12.38) | 67.8 (7.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 19 | 22 | 2 | 63
  Male | 17 | 18 | 12 | 2 | 49
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 1
  Asian | 0 | 3 | 1 | 0 | 4
  Black or African American | 0 | 1 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  White | 35 | 31 | 32 | 4 | 102
  Other | 2 | 1 | 0 | 0 | 3
  Unknown | 0 | 0 | 0 | 0 | 0
  Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Canada | 7 | 6 | 7 | 0 | 20
  United Kingdom | 10 | 10 | 13 | 0 | 33
  Australia | 20 | 21 | 14 | 4 | 59
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m2] | 30.39 (4.473) | 31.20 (5.131) | 33.01 (5.185) | 29.58 (1.431) | 31.42 (4.934)

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve (AUC) for the Numeric Rating Scale at Rest (NRS-R) of Pain Intensity.
Description: NRS-R for pain intensity is an 11-item scale from 0 to10 where participants rank the level of pain intensity. The NRS scale goes from No Pain (0) to Worst Imaginable Pain (10).
Time Frame: from 30 minutes post-surgery through hour 168 (Day 8)
Population: Full analysis set (FAS)
Measure: Mean (Standard Deviation); unit: pain intensity score*hour
Arm/Group | ATX-101 1000 mg | ATX-101 1500 mg | Bupivacaine Hydrochloride | Saline Placebo
Number analyzed (Participants) | 37 | 37 | 34 | 4
pain intensity score*hour | 517.32 (284.675) | 518.03 (239.299) | 595.26 (258.945) | 756.84 (261.454)

2. Secondary Outcome: Percentage of Subject Who Remain Opioid Free.
Description: Opioid free is defined as no opioid rescue medication was recorded for the timepoint displayed and onwards.
Time Frame: Surgical Closure to Day 30
Population: Full Analysis Set (FAS)
Measure: Count of Participants; unit: Participants
Arm/Group | ATX-101 1000 mg | ATX-101 1500 mg | Bupivacaine Hydrochloride | Saline Placebo
Number analyzed (Participants) | 37 | 37 | 34 | 4
Participants
  Surgical Closure - Day 30 | 3 | 6 | 1 | 0
  Day 4 - Day 30 | 12 | 13 | 6 | 0
  Day 5 - Day 30 | 13 | 15 | 6 | 0
  Day 8 - Day 30 | 14 | 17 | 10 | 1
  Day 15 - Day 30 | 17 | 22 | 16 | 1
  Day 22 - Day 30 | 24 | 27 | 23 | 1

3. Secondary Outcome: Total Post-surgical Use of Rescue Opioid Medications.
Description: Total post-surgical use of rescue opioid medications (days).
Time Frame: Surgical Closure to Day 30, Opioid consumption is summarized descriptively every 24-hour period through Day 30
Population: Full Analysis Set (FAS)
Measure: Mean (Standard Deviation); unit: IV Morphine Milligram Equivalent (MME)
Arm/Group | ATX-101 1000 mg | ATX-101 1500 mg | Bupivacaine Hydrochloride | Saline Placebo
Number analyzed (Participants) | 37 | 37 | 34 | 4
IV Morphine Milligram Equivalent (MME)
  Surgical Closure - Hour 24 (Day 1): number analyzed (Participants) | 31 | 29 | 30 | 4
  Surgical Closure - Hour 24 (Day 1) | 63.153 (62.6833) | 58.399 (47.1712) | 43.283 (29.0513) | 119.800 (58.1316)
  Hour 24 (Day 1) - Hour 48 (Day 2): number analyzed (Participants) | 29 | 28 | 28 | 4
  Hour 24 (Day 1) - Hour 48 (Day 2) | 44.628 (40.0835) | 33.566 (29.9608) | 36.804 (30.9289) | 107.250 (50.5486)
  Hour 48 (Day 2) - Hour 72 (Day 3): number analyzed (Participants) | 20 | 22 | 20 | 3
  Hour 48 (Day 2) - Hour 72 (Day 3) | 30.500 (25.1244) | 25.795 (18.9251) | 32.550 (21.3338) | 40.000 (8.6603)
  Hour 72 (Day 3) - Day 4: number analyzed (Participants) | 17 | 15 | 21 | 3
  Hour 72 (Day 3) - Day 4 | 24.044 (22.3062) | 23.783 (19.7504) | 25.369 (16.9465) | 35.000 (22.9129)
  Day 4 - Day 5: number analyzed (Participants) | 15 | 14 | 17 | 3
  Day 4 - Day 5 | 26.733 (26.0054) | 22.214 (18.1274) | 23.853 (20.0357) | 37.500 (19.8431)
  Day 5 - Day 6: number analyzed (Participants) | 14 | 16 | 15 | 3
  Day 5 - Day 6 | 25.000 (21.5058) | 24.063 (22.5092) | 25.067 (25.0933) | 40.000 (22.9129)
  Day 6 - Day 7: number analyzed (Participants) | 17 | 13 | 20 | 3
  Day 6 - Day 7 | 27.206 (21.8818) | 18.923 (13.2725) | 26.225 (21.1209) | 27.500 (15.6125)
  Day 7 - Day 8: number analyzed (Participants) | 17 | 14 | 16 | 3
  Day 7 - Day 8 | 19.147 (13.7509) | 16.000 (9.7033) | 28.219 (20.8734) | 18.750 (9.9216)
  Day 8 - Day 9: number analyzed (Participants) | 17 | 12 | 15 | 3
  Day 8 - Day 9 | 19.147 (10.3089) | 21.042 (17.0140) | 19.833 (13.7369) | 25.000 (17.3205)
  Day 9 - Day 10: number analyzed (Participants) | 17 | 11 | 13 | 3
  Day 9 - Day 10 | 20.176 (13.4768) | 15.045 (8.3260) | 20.192 (13.8241) | 20.000 (11.4564)
  Day 10 - Day 11: number analyzed (Participants) | 14 | 11 | 15 | 2
  Day 10 - Day 11 | 20.214 (12.4216) | 17.591 (10.9654) | 21.100 (13.8824) | 12.750 (3.1820)
  Day 11 - Day 12: number analyzed (Participants) | 15 | 12 | 14 | 3
  Day 11 - Day 12 | 16.417 (12.7201) | 14.208 (11.3367) | 15.875 (8.0770) | 15.000 (7.5000)
  Day 12 - Day 13: number analyzed (Participants) | 14 | 10 | 15 | 3
  Day 12 - Day 13 | 16.071 (10.7289) | 15.900 (9.1767) | 21.567 (14.9354) | 12.500 (4.3301)
  Day 13 - Day 14: number analyzed (Participants) | 14 | 11 | 15 | 1
  Day 13 - Day 14 | 13.571 (7.1195) | 14.591 (7.5459) | 19.500 (12.8504) | 30.000 (NA) — standard deviation cannot be calculated for one participant
  Day 14 - Day 15: number analyzed (Participants) | 15 | 10 | 11 | 2
  Day 14 - Day 15 | 20.200 (17.2293) | 13.850 (9.6149) | 14.091 (6.5453) | 15.000 (10.6066)
  Day 15 - Day 16: number analyzed (Participants) | 11 | 7 | 14 | 2
  Day 15 - Day 16 | 17.045 (11.6092) | 17.571 (7.7051) | 12.321 (8.5605) | 15.000 (10.6066)
  Day 16 - Day 17: number analyzed (Participants) | 14 | 9 | 11 | 2
  Day 16 - Day 17 | 14.821 (7.8117) | 11.167 (4.1307) | 18.682 (10.6941) | 15.000 (10.6066)
  Day 17 - Day 18: number analyzed (Participants) | 12 | 10 | 11 | 2
  Day 17 - Day 18 | 14.271 (8.7331) | 12.700 (5.7359) | 10.232 (8.8154) | 15.000 (10.6066)
  Day 18 - Day 19: number analyzed (Participants) | 13 | 4 | 14 | 3
  Day 18 - Day 19 | 17.981 (20.5113) | 12.500 (6.1237) | 11.411 (9.1744) | 7.500 (0.0000)
  Day 19 - Day 20: number analyzed (Participants) | 10 | 4 | 9 | 2
  Day 19 - Day 20 | 17.550 (14.2993) | 7.875 (0.7500) | 14.722 (10.1122) | 11.250 (5.3033)
  Day 20 - Day 21: number analyzed (Participants) | 9 | 7 | 8 | 2
  Day 20 - Day 21 | 17.778 (15.1783) | 13.000 (9.5481) | 12.563 (5.2809) | 7.500 (0.0000)
  Day 21 - Day 22: number analyzed (Participants) | 11 | 6 | 9 | 3
  Day 21 - Day 22 | 17.273 (14.3267) | 11.083 (5.5083) | 10.972 (4.9124) | 7.500 (0.0000)
  Day 22 - Day 23: number analyzed (Participants) | 9 | 4 | 6 | 3
  Day 22 - Day 23 | 19.861 (17.0069) | 9.750 (3.5707) | 13.750 (5.6458) | 18.333 (18.7639)
  Day 23 - Day 24: number analyzed (Participants) | 10 | 5 | 6 | 3
  Day 23 - Day 24 | 16.750 (14.1323) | 11.000 (4.1683) | 11.250 (4.1079) | 31.667 (41.8579)
  Day 24 - Day 25: number analyzed (Participants) | 8 | 5 | 6 | 3
  Day 24 - Day 25 | 13.906 (14.7515) | 13.400 (11.0872) | 13.750 (3.0619) | 18.333 (18.7639)
  Day 25 - Day 26: number analyzed (Participants) | 7 | 7 | 5 | 2
  Day 25 - Day 26 | 18.750 (14.2705) | 12.357 (9.0725) | 13.500 (3.3541) | 7.500 (0.0000)
  Day 26 - Day 27: number analyzed (Participants) | 8 | 7 | 5 | 2
  Day 26 - Day 27 | 9.844 (6.1397) | 9.857 (3.8699) | 11.250 (7.5000) | 23.750 (22.9810)
  Day 27 - Day 28: number analyzed (Participants) | 5 | 5 | 3 | 0
  Day 27 - Day 28 | 18.500 (20.6610) | 12.700 (6.9964) | 10.000 (4.3301) |
  Day 28 - Day 29: number analyzed (Participants) | 6 | 5 | 4 | 1
  Day 28 - Day 29 | 17.917 (19.1974) | 11.700 (5.9224) | 6.563 (1.8750) | 20.000 (NA) — standard deviation cannot be calculated for one participant
  Day 29 - Day 30: number analyzed (Participants) | 1 | 1 | 2 | 0
  Day 29 - Day 30 | 47.500 (NA) — standard deviation cannot be calculated for one participant | 16.000 (NA) — standard deviation cannot be calculated for one participant | 7.500 (0.0000) |

4. Secondary Outcome: Time to First Rescue Opioid Medication.
Description: Time to first postsurgical use of rescue opioid medication (days).
Time Frame: Surgical Closure to Day 30
Population: Full Analysis Set (FAS)
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | ATX-101 1000 mg | ATX-101 1500 mg | Bupivacaine Hydrochloride | Saline Placebo
Number analyzed (Participants) | 37 | 37 | 34 | 4
Days | 0.478 (0.9862) | 0.257 (0.2571) | 0.491 (0.6925) | 0.223 (0.0820)

ADVERSE EVENTS:
Time Frame: Day 56
Description: AEs were collected from the time of the investigational product administration and followed until the resolution of AE(s) or the Day 56 Visit, whichever occurred first.
Arm/Group | ATX-101 1000 mg | ATX-101 1500 mg | Bupivacaine Hydrochloride | Saline Placebo
All-Cause Mortality (participants affected / at risk) | 0/37 | 0/37 | 0/34 | 0/4
Serious Adverse Events (participants affected / at risk) | 3/37 | 4/37 | 2/34 | 0/4
Other Adverse Events (participants affected / at risk) | 30/37 | 25/37 | 28/34 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ATX-101 1000 mg (N=37) | ATX-101 1500 mg (N=37) | Bupivacaine Hydrochloride (N=34) | Saline Placebo (N=4)
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Liver injury (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Incision site discharge (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 1 | 0 | 0
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Delirium (Psychiatric disorders) | 0 | 1 | 0 | 0
Pulmonary embolism (Vascular disorders) | 0 | 1 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ATX-101 1000 mg (N=37) | ATX-101 1500 mg (N=37) | Bupivacaine Hydrochloride (N=34) | Saline Placebo (N=4)
Constipation (Gastrointestinal disorders) | 5 | 4 | 9 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 2 | 1 | 0
Nausea (Gastrointestinal disorders) | 11 | 10 | 9 | 2
Procedural pain (Injury, poisoning and procedural complications) | 2 | 4 | 5 | 0
Contusion (Injury, poisoning and procedural complications) | 3 | 2 | 4 | 0
Dizziness (Nervous system disorders) | 3 | 6 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 2 | 4 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 1 | 2 | 0
Vomiting (Gastrointestinal disorders) | 3 | 0 | 4 | 0
Implant site swelling (General disorders) | 1 | 3 | 2 | 0 — General disorders and administration site conditions
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 2 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Material for public dissemination will be submitted to the Sponsor for review at least sixty (60) days (or the time specified in the Protocol if longer) prior to submission for publication, public dissemination, or review by a publication committee. Principal Investigator agrees that all reasonable comments made by the Sponsor in relation to a proposed publication by the Trial Site, any Other Trial Site, and/or the Principal Investigator will be incorporated into the publication.

DOCUMENTS (2):
  • Study Protocol (2023-06-02): https://cdn.clinicaltrials.gov/large-docs/08/NCT05260008/Prot_000.pdf
  • Statistical Analysis Plan (2024-02-20): https://cdn.clinicaltrials.gov/large-docs/08/NCT05260008/SAP_001.pdf